CLINICAL TRIAL: NCT00001729
Title: Combination of Alpha Interferon With Long Term Ribavirin Therapy for Patients With Chronic Hepatitis C
Brief Title: Combination Drug Therapy for Patients With Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980003; 98-DK-0003
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-09

CONDITIONS: Chronic Hepatitis C; Fibrosis; Hemolytic Anemia
Keywords: Cirrhosis; Liver Disease; Hemolytic Anemia; Liver Biopsy; Ribavirin; Alpha Interferon; Viral Hepatitis; Hepatitis C Virus; Chronic Hepatitis; Antiviral Agents
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis; Anemia, Hemolytic; Liver Diseases; Hepatitis C; Hepatitis, Chronic | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirin

SUMMARY:
Hepatitis C is a major cause of liver disease in the United States and leads to cirrhosis of the liver in approximately one-third of patients some of whom will ultimately suffer from liver failure or liver cancer. At present, the recommended therapy of hepatitis C is the combination of alpha interferon and ribavirin given for 6 to 12 months. Ribavirin is a antiviral drug that is given by mouth. Interferon is both an antiviral and an immune medication which must be given by injections (three times a week) and has many difficult side effects. The purpose of this study is to determine whether the combination of ribavirin and interferon improve the liver disease of hepatitis C and whether improvements can be maintained by continuing ribavirin therapy long-term. This study will take 100 to 120 patients suffering from hepatitis C and place them under combination drug therapy with alpha interferon and ribavirin. The course of drug therapy is scheduled to last 6 to 12 months. Patients will be selected after appropriate screening for hepatitis C virus and elevated liver enzymes are conducted and liver biopsy shows chronic hepatitis with some degree of injury and scarring.

During the first 6 months of the study, subjects will be asked to return to the outpatient clinic for routine check-ups and blood tests every 2 to 4 weeks. Blood tests will include tests for hepatitis C virus. If the virus test becomes negative on treatment, the therapy will be considered successful and will be continued for a full 6 or 12 months (depending upon the strain of virus).

If the virus test does not become negative during the first six months of treatment, subjects will be considered "non-responders" and will stop taking interferon but will continue on ribavirin alone or an identically appearing placebo tablet. These non-responsive subjects will continue this therapy for an additional 12 months. (A year-and-a-half total).

Upon completion of the drug therapies, subjects will be requested to submit blood samples and undergo a liver biopsy to determine if the therapy was successful. Test results that reveal a loss of hepatitis C antibodies or normal levels of liver enzymes will be deemed successful.

Patients that have successful laboratory test results will be considered for continuation of ribavirin therapy. Patients that received placebo for a year will be eligible to receive ribavirin long-term at the end of the study.

DETAILED DESCRIPTION:
Between 60 and 90 patients with chronic hepatitis C will be enrolled in a study of the combination of alpha interferon and ribavirin for 12 months with early discontinuation of therapy and randomization to receive either ribavirin alone or placebo for patients who do not respond within 6 months of starting therapy. Adult patients will be chosen who have chronic hepatitis C, HCV RNA in serum, and elevations in serum aminotransferases. Patients who have received alpha interferon in the past will be eligible if they did not have a sustained response to their previous course of interferon. After medical evaluation and liver biopsy, patients will begin receiving alpha interferon by subcutaneous injection in a dose of 3 million units three times weekly. At the same time, patients will begin receiving ribavirin orally in a dose of 1000 mg (if body weight is less than 75 kg) or 1200 mg daily (two or three capsules of 200 mg twice daily). During the initial 24-week period of combination therapy, patients will be seen in the outpatient clinic for medical interview, physical examinations and blood tests at 2 to 4 week intervals. At 24 weeks, patients will be classified as either responders or non-responders based upon HCV RNA testing of serum. Responders will continue on the combination therapy for another 24 weeks (total treatment = 48 weeks). Non-responders will stop interferon therapy and will be randomized to receive either ribavirin or identically appearing placebo capsules for 48 weeks (total treatment = 72 weeks). At the 72 week point (18 months after enrollment), all patients will be readmitted for repeat medical evaluation and liver biopsy. At this point, ribavirin and placebo will be stopped (unless the patient has had a clear histological and biochemical response to therapy) and patients will be monitored with outpatient visits at 8 week intervals for another 6 months.

Patients who exhibit a histological and biochemical response to ribavirin monotherapy will be offered a one-year extension of treatment with ribavirin in a gradually reduced dosage. These patients will be monitored at 8 week intervals and the dose will be reduced by 200 mg per day every 16 weeks to a minimum dose of 600 mg per day. If the biochemical response is maintained, patients will continue on therapy for one year and then undergo repeat medical evaluation and liver biopsy. Continued therapy with ribavirin after this point will depend upon whether safety and efficacy of ribavirin have been demonstrated and whether ribavirin has been approved for use in hepatitis C.

The primary criterion for success of therapy overall will be sustained loss of HCV RNA as assessed at 18 months. Primary criteria for response among the patients who are randomized to receive ribavirin or placebo will be degree of histological improvement on liver biopsy. Secondary criteria will be normalization of ALT levels. This study will allow for therapy of all patients with chronic hepatitis C with the combination of alpha interferon and ribavirin and will allow for therapy of patients with resistant forms of chronic hepatitis C with ribavirin alone and will address whether monotherapy with ribavirin can sustain these improvements and whether the biochemical improvements reflect amelioration of the underlying liver disease as judged histologically.

ELIGIBILITY:
INCLUSION CRITERIA:

Age above 18 years, male or female.

Serum alanine or asparate aminotransferase activities that are above the upper limit of normal (ALT greater than 41 or AST greater than 31 U/L) on an average of three determinations taken during the previous 6 months. The mean of the three determinations will be defined as "baseline" levels.

Presence of anti-HCV and HCV RNA in serum tested at least once during the previous six months.

Evidence of chronic hepatitis on liver biopsy done within the previous 12 months with a histology activity index of at least 6 (out of a maximum of 22).

Written informed consent.

EXCLUSION CRITERIA:

If previously treated with interferon or ribavirin, must not have a lack of sustained virological response as shown by the presence of HCV RNA in serum six months after stopping therapy. Patients must not have received the combination of alpha interferon and ribavirin in the past.

Decompensated liver disease, as marked by bilirubin greater than 4 mg%, albumin less than 3.0 gm%, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Patients with ALT levels greater than 1000 U/L (greater than 25 times ULN) will not be enrolled but may be followed until three determinations are below this level.

Pregnancy or, in women of child-bearing potential or spouses of such women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermacide, or birth control pills, or an intrauterine device.

Significant systemic or major illnesses other than liver disease, including congestive heart failure, renal failure (creatinine clearance less than 50 ml/min), organ transplantation, serious psychiatric disease or depression, and angina pectoris.

Pre-existing anemia (hematocrit less than 36% for men and less than 34% for women) or known history of hemolytic anemia.

Antiviral or immunosuppressive therapy within the last 6 months.

Evidence of another form of liver disease in addition to viral hepatitis (e.g., autoimmune liver disease, Wilson's disease, alcoholic liver disease, hemochromatosis, alpha-1-antitrypsin deficiency).

Any evidence of coronary artery disease or cerebral vascular disease, including abnormalities on exercise stress testing in patients with defined risk factors who will be screened for evidence of underlying coronary artery disease.

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.

Evidence of hepatocellular carcinoma; either alphafetoprotein (AFP) levels greater than 50 ng/ml (normal is less than 9 ng/ml) and /or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.

Clinical gout.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1997-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Alter HJ. Descartes before the horse: I clone, therefore I am: the hepatitis C virus in current perspective. Ann Intern Med. 1991 Oct 15;115(8):644-9. doi: 10.7326/0003-4819-115-8-644. PMID 1654040
- [Background] Major ME, Feinstone SM. The molecular virology of hepatitis C. Hepatology. 1997 Jun;25(6):1527-38. doi: 10.1002/hep.510250637. No abstract available. PMID 9185778
- [Background] Kiyosawa K, Sodeyama T, Tanaka E, Gibo Y, Yoshizawa K, Nakano Y, Furuta S, Akahane Y, Nishioka K, Purcell RH, et al. Interrelationship of blood transfusion, non-A, non-B hepatitis and hepatocellular carcinoma: analysis by detection of antibody to hepatitis C virus. Hepatology. 1990 Oct;12(4 Pt 1):671-5. doi: 10.1002/hep.1840120409. PMID 2170265